CLINICAL TRIAL: NCT01938404
Title: Post-Marketing Requirement Study to Evaluate the Safety and Efficacy of Octaplas™ in Patients With Thrombotic Thrombocytopenic Purpura With Special Emphasis on Monitoring the Occurrence of Thromboembolic Events
Brief Title: Octaplas Adult TTP Trial
Status: Terminated | Type: Observational
Why Stopped: FDA released from conducting
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: LAS-214
Record Dates: First submitted 2013-09-02; First posted 2013-09-10 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: Plasma exchange; Thrombotic Thrombocytopenic Purpura; TTP
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Octaplas: Patients receiving Octaplas for the treatment of Thrombotic Thrombocytopenic Purpura (TTP) undergoing therapeutic plasma exchange (TPE) procedures
  Interventions: Biological: Octaplas
- standard plasma products: Patients receiving standard plasma products (e.g., FFP, etc) for the treatment of Thrombotic Thrombocytopenic Purpura (TTP) undergoing therapeutic plasma exchange (TPE) procedures
  Interventions: Drug: Standard Plasma

INTERVENTIONS:
Biological: Octaplas — Octoplas infusion solution for IV administration
  Groups: Octaplas
Drug: Standard Plasma — Plasma given as replacement fluid
  Other Names: FFP, FP24, 5 day plasma
  Groups: standard plasma products

SUMMARY:
To assess and evaluate the safety of octaplas™ in comparison to standard plasma product (e.g., fresh frozen plasma (FFP) and other approved plasma products used within 24 hours of thawing) used in the treatment of TTP, in patients undergoing Therapeutic Plasma Exchange, with a special emphasis on the occurrence of thromboembolic events (TEEs).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or female at least 18 years of age or older.
2. Patient has a diagnosis of TTP or suspicion of TTP that is planned on being treated with TPE within 3 days of study entry.
3. Patient has thrombocytopenia (platelets < 100 x 10P9P/L).
4. Patient is willing to give voluntary written informed consent before any study-related procedure is to be performed that is not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Patient has a history of severe hypersensitivity reaction to plasma-derived products or to FFP.
2. Patient has an already known IgA deficiency with documented antibodies against IgA.
3. Patient is currently participating in an interventional clinical study or has participated during the past 1 month prior to study inclusion.
4. Patient has severe deficiencies of Protein S.
5. Patient received more than 1 treatment of plasma exchange or plasma infusion for current episode of TTP prior to randomization.
6. Patient is currently taking ACE-inhibitors; in case patient is under ACE-inhibitor treatment a wash-out period of at least 24 hours has to elapse prior the first plasma infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing Plasma exchange for Thrombotic Thrombocytopenic Purpura
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
The incidence of TEEs in patients receiving octaplas™ will be compared with the incidence rate in patients receiving plasma issued according to institutional standard of care. | Up to 28 days followed by a 24 hour follow-up

SECONDARY OUTCOMES:
Incidence of Citrate reactions during TPE based on clinical judgment of physician. | Up to 28 days followed by a 24 hour follow-up
Incidence of Plasma-associated adverse reactions including Transfusion-Associated Circulatory Overload (TACO), | Up to 28 days followed by a 24 hour follow-up
Incidence of Transfusion-Related Acute Lung Injury (TRALI) | Up to 28 days followed by a 24 hour follow-up
Incidence of febrile reactions | Up to 28 days followed by a 24 hour follow-up
Measurement of Safety laboratory parameters - International Normalized Ratio (INR) | Up to 28 days followed by a 24 hour follow-up
Measurement of Prothrombin Time (PT)/Partial Thromboplastin Time (PTT). | Up to 28 days followed by a 24 hour follow-up
Determination of overall clinical response (rating scale that takes into account platelet count, LDH levels, creatinine and neurological status). | Up to 28 days followed by a 24 hour follow-up
measurement of Platelet count | Up to 28 days followed by a 24 hour follow-up
measurement of hemoglobin | Up to 28 days followed by a 24 hour follow-up
measurement of hematocrit | Up to 28 days followed by a 24 hour follow-up
measurement of LDH. | Up to 28 days followed by a 24 hour follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Study Director — International Medical Director
Locations (2):
- United States (2):
  - Octapharma Study Site, Manhasset, New York
  - Octapharma Study Site, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes